CLINICAL TRIAL: NCT01765127
Title: An Observational Post-Authorization Modified Prescription-Event Monitoring Safety Study to Monitor the Safety and Utilization of Asenapine (Sycrest) in the Primary Care Setting in England
Brief Title: An Observational Modified Prescription-event Monitoring Study of Asenapine (Sycrest)
Status: Completed | Type: Observational
Sponsor: Professor Saad Shakir (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Professor Saad Shakir, Director, Drug Safety Research Unit, Southampton, UK
Organization: Drug Safety Research Unit, Southampton, UK (Other)
Other Study IDs: Asenapine ModPEM
Record Dates: First submitted 2012-12-18; First posted 2013-01-10 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Bipolar I Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asenapine: Patients prescribed asenapine for any indication by a National Health Service (NHS) general practitioner (GP) in England.

SUMMARY:
This post-marketing Modified Prescription-Event Monitoring (M-PEM) safety study of asenapine (SYCREST®) is to be carried out by the Drug Safety Research Unit (DSRU) as part of the Risk Management Plan required by the Committee for Medicinal Products for Human Use (CHMP) to further investigate the safety profile of asenapine in clinical practice. The aim of this study is to proactively capture safety and drug utilisation data in the post-marketing phase of license approval of asenapine as prescribed to patients by general practitioners (GPs) in England. This data is obtained through the completion of questionnaires by GPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed asenapine for any indication by NHS GPs in England.
* Patients for whom a study questionnaire containing useful information has been returned, will be included in the study cohort regardless of the dose or frequency of administration of asenapine, and irrespective of whether any medicines are concurrently administered.

Exclusion Criteria:

* patient no longer registered with the practice
* patient for whom no information is provided on study questionnaire
* patients for whom information provided on study questionnaire relates to another antipsychotic drug
* patients for whom the index date is an improbable date (i.e. before market launch date)
* patients for whom the GP reports that the patient did not take or was never prescribed asenapine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients prescribed asenapine for any indication by NHS GPs in England.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2012-01; Primary Completion 2017-02 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of selected important identified and potential risks | At least 3 months after drug is first prescribed.
  Incidence rates of these risks will be quantified:
  * Somnolence and sedation
  * Weight gain
  * Oral hypoaesthesia
  * Swelling of the tongue and throat
  * Allergic reactions (Type 1 hypersensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Shakir, Professor, Principal Investigator — Drug Safety Research Unit
Locations (1):
- Drug Safety Research Unit (for data collation and analysis only), Southampton, Hampshire, United Kingdom